CLINICAL TRIAL: NCT07015996
Title: Efficacy of Tezepelumab in Peanut Oral Immunotherapy: a Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: Efficacy of Tezepelumab in Peanut Oral Immunotherapy
Acronym: ZENITH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ITN097AD
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Peanut Allergy
Keywords: Tezepelumab; Peanut; Oral Immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab plus Peanut Oral Immunotherapy (OIT) Group (Experimental): Eligible participants will be randomized in a 1:1 fashion to receive Tezepelumab during the monotherapy period of the trial. Throughout the combination therapy period, which also includes an OIT build-up and maintenance period, participants will remain on tezepelumab 210 mg every 4 weeks until reaching the final period of the trial, the withdrawal period.
  Interventions: Biological: Tezepelumab; Drug: Peanut Oral Immunotherapy (OIT)
- Placebo for Tezepelumab plus peanut Oral Immunotherapy (OIT) Group (Placebo Comparator): Eligible participants will be randomized in a 1:1 fashion to receive placebo for Tezepelumab during the monotherapy period of the trial. Throughout the combination therapy period, which also includes an OIT build-up and maintenance period, participants will remain on placebo for tezepelumab every 4 weeks until reaching the final period of the trial, the withdrawal period.
  Interventions: Drug: Peanut Oral Immunotherapy (OIT); Biological: Placebo for Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — Monotherapy Period: Participants randomized to tezepelumab will receive two subcutaneous (SQ) injections of tezepelumab 210 mg during the monotherapy period.
  Combination Therapy Period: Participants randomized to Tezepelumab will continue to receive Tezepelumab 210 mg every 4 weeks.
  Withdrawal Period: Participants will stop receiving Tezepelumab injections.
  Arms: Tezepelumab plus Peanut Oral Immunotherapy (OIT) Group
Drug: Peanut Oral Immunotherapy (OIT) — Monotherapy Period: Not Applicable. Combination Therapy Period: During combination therapy period, each participant will start peanut OIT. Participants will start on a minimum of 0.1 mg peanut OIT, with starting dose depending on last tolerated dose from screening double-blind placebo-controlled food challenge (DBPCFC) and build to a maximum of 6 mg peanut OIT on the initial dose escalation (IDE) day. Participants will return every 2 weeks for dose escalation to a goal maintenance dose of 2000 mg peanut protein.
  Withdrawal Period: Participants will stop peanut OIT.
Biological: Placebo for Tezepelumab — Monotherapy Period: Participants randomized to placebo for tezepelumab will receive two subcutaneous (SQ) injections of placebo 210 mg during the monotherapy period.
  Combination Therapy Period: Participants randomized to placebo will continue to receive placebo for Tezepelumab every 4 weeks.
  Withdrawal Period: Participants will stop receiving placebo injections.
  Arms: Placebo for Tezepelumab plus peanut Oral Immunotherapy (OIT) Group

SUMMARY:
The proposed study is a proof-of-concept Phase 2, double-blind, randomized placebo-controlled clinical trial evaluating the safety and efficacy of tezepelumab and peanut Oral Immunotherapy (OIT) for the treatment of peanut allergy. Study participation is divided into 3 periods: (i) a monotherapy period comprised of injections of either Tezepelumab or placebo from week 0 to week 8, (ii) followed by a combination therapy period comprised of 56 weeks during which peanut OIT is built up and maintained, and (iii) a treatment withdrawal period comprised of 12 weeks. This study will enroll 62 peanut-allergic individuals from 12 to 55 years of age who experience dose-limiting symptoms to <=100 mg of peanut protein in a single dose (<= 144 mg cumulative dose) as assessed by DBPCFC.

The primary objective is to determine whether 56 weeks of tezepelumab plus peanut OIT as compared to 56 weeks of placebo plus peanut OIT induces sustained unresponsiveness to peanut 12 weeks after stopping combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent/legal guardian must be able to understand and provide informed consent (parental permission and informed assent of minor, if applicable)
2. A personal history of an allergic reaction to peanut ingestion
3. A positive reaction at or below ingestion of 100 mg of peanut protein in a single dose (<= 144 milligram cumulative dose) during the screening Double-Blind Placebo-Controlled Food Challenge (DBPCFC)
4. A negative challenge to the placebo (oat) during the Screening DBPCFC
5. Sensitization to peanut as evidenced by either one of the following:

   1. positive sIgE to Ara h2 >= 0.35 kilounit per liter by ImmunoCAP (TM) testing, or
   2. wheal >= 3 mm on skin prick test to peanut extract compared to a negative control
6. Female participants of childbearing potential must have a negative pregnancy test upon study entry
7. Female participants with reproductive potential must agree to use an FDA approved method of contraception for the duration of the study
8. Willing and able to comply with the study protocol requirements
9. Participants with other food allergies must agree to continue avoidance of these food items from their diet to avoid confounding the safety and efficacy data of the study

Exclusion Criteria:

1. Currently in build-up phase of aeroallergen immunotherapy
2. Current food allergen immunotherapy or use of any food allergen immunotherapy within the past 12 months
3. Pregnant, planning a pregnancy during the study, or breast-feeding
4. History of intolerance, hypersensitivity, or allergic reactions to tezepelumab, or the inactive ingredients (excipients) of tezepelumab, other IgG biologics, or rescue medications and their excipients
5. Allergy to oat (participant reported)
6. History of severe systemic allergic reaction to peanut with symptoms including the need for mechanical ventilation and/or severe hypotension requiring intensive care unit admission
7. Asthma requiring high dose inhaled corticosteroid therapy for control (2007 NHLBI Criteria Steps 5 or 6 in adults and adolescents)
8. History of a life-threatening asthma attack within 1 year before screening (e.g., requiring an ICU admission or intubation with mechanical ventilation), need for oral corticosteroids for asthma management within the last 6 months, or current Asthma Control Test score less than 19 at screening
9. History of ischemic cardiovascular disease or other cardiac disease, where, in the opinion of the site investigator, participation in the trial would pose a risk from participation in the study
10. History of eosinophilic gastrointestinal disease at screening
11. History of disease affecting the immune system such as autoimmune disease (e.g., systemic lupus erythematosus), immune complex disease (e.g., serum sickness), or immunodeficiency, where, in the opinion of the site investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
12. History of malignancy of any type, excluding basal cell and squamous cell cancers of the skin that only required surgical excision or in situ carcinoma of the cervix study provided that curative therapy was completed at least 12 months prior to informed consent
13. Current known helminth infection
14. Positive QuantiFERON - TB Gold test or TB Gold Plus, or T-SPOT(R) TB test unless the potential participant has been treated with appropriate chemoprophylaxis. In the case of an indeterminate or borderline Interferon Gamma Release Assay (IGRA), an IGRA may be repeated
15. Any of the following:

    1. HIV
    2. current or prior infection with hepatitis B virus (HBV)
    3. current or prior infection with hepatitis C virus (HCV), except adequately treated HCV with sustained virologic response >= 12 weeks
16. Active liver disease, defined as either:

    1. AST, ALT, and/or Alk phos >2x ULN, or
    2. other active liver disease which, in the opinion of the site investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
17. Any of the following:

    1. Current use of beta-blockers, angiotensin-converting enzyme inhibitors, or angiotensin-receptor blockers
    2. Received any investigational product within the past 4 months or 5 half-lives (whichever is longer) prior to screening
    3. Received systemic corticosteroids within 14 days prior to screening
    4. Receipt of immunoglobulin or other blood product within 30 days of screening
    5. Receipt of live attenuated vaccine within 30 days of informed consent
    6. Use of an immunosuppressant or immunomodulating drug within 30 days prior to screening
    7. Use of biologics targeting the human immune system within the past 12 months prior to screening
    8. Use of any herbal medications, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
18. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the site investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02-18 (Estimated); Primary Completion 2028-09-16 (Estimated); Study Completion 2028-09-16 (Estimated)

PRIMARY OUTCOMES:
Consumption of a cumulative dose of 4000 mg of peanut protein without dose-limiting symptoms during the open Oral Food Challenge (OFC) | At week 76
  The primary endpoint is sustained unresponsiveness to peanut 12 weeks after stopping combination therapy, as assessed by passing the open OFC to peanut at Week 76

SECONDARY OUTCOMES:
Highest single dose of peanut protein consumed without doselimiting symptoms during the open Oral Food Challenge (OFC) | At week 64 and 76
Consumption of a cumulative dose of 4000 mg of peanut protein without doselimiting symptoms during the open Oral Food Challenge (OFC) | At week 64
Highest cumulative dose of peanut protein consumed without dose limiting symptoms during the open Oral Food Challenge (OFC) | At week 64 and 76
An adverse event related to monotherapy | During 8 weeks of therapy
An adverse event related to combination therapy | During 56 weeks of therapy
An adverse event related to tezepelumab plus peanut Oral Immunotherapy (OIT) discontinuation | 12 weeks after discontinuation of treatment
An adverse event related to placebo plus peanut Oral Immunotherapy (OIT) discontinuation | 12 weeks after discontinuation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edwin H Kim, M.D., M.S., Study Chair — North Carolina Children's Hospital: Department of Pediatrics, Division of Allergy, Immunology and Rheumatology; Sarita Patil, M.D., Study Chair — Massachusetts General Hospital: Department of Medicine: Allergy & Clinical Immunology Unit
Locations (10):
- United States (10):
  - Arkansas Children's Hospital Research Institute: Department of Pediatrics, Allergy & Immunology, Little Rock, Arkansas
  - University of California, Los Angeles: Department of Medicine, Division of Clinical Immunology and Allergy, Los Angeles, California
  - Johns Hopkins Children's Center: Department of Allergy & Immunology, Baltimore, Maryland
  - Massachusetts General Hospital: Department of Medicine: Allergy & Clinical Immunology Unit, Boston, Massachusetts
  - Boston Children's Hospital: Allergy and Asthma Program, Boston, Massachusetts
  - The University of Michigan: Division of Allergy and Clinical Immunology, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai: Department of Pediatrics Allergy & Immunology, New York, New York
  - North Carolina Children's Hospital: Department of Pediatrics, Division of Allergy, Immunology and Rheumatology, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center: Division of Allergy and Immunology, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center: Division of Allergy and Immunology, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: http://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait